CLINICAL TRIAL: NCT03412617
Title: Association of Intake and Nutritional Status With Total Microbiota and Metabolic Marker in Minangkabau and Sundanese Women in Urban and City: A Comparative Study
Brief Title: Diets, Metabolic Profile and Gut Microbiota Among Indonesian Women in Minangkabau and Sundanese-ethnic Community
Status: Completed | Type: Observational
Sponsor: Rina Agustina (Other)
Collaborators: SEAMEO Regional Centre for Food and Nutrition (Other); Indonesia University (Other)
Responsible Party: Sponsor-Investigator, Rina Agustina, MD, MSc, PhD, Indonesia University
Organization: Indonesia University (Other)
Other Study IDs: Dietary Minangkabau-Sunda
Record Dates: First submitted 2018-01-11; First posted 2018-01-26 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Healthy Women; Diet Habit; Bifidobacterium; Inflammation; Obesity; Blood Glucose, High
Keywords: Healthy Eating; Blood glucose; Bifidobacterium; Obese women
MeSH Terms: conditions — Feeding Behavior; Inflammation; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many provinces in Indonesia have some well known traditional foods that are widely consumed, but it remains unknown whether traditional ethnic dietary patterns can confirm healthy diets. High quality diet is associated with reduced risk of metabolic diseases and modulated gut microbiota. Moreover, the relationship between dietary quality and microbiota, a potential mediator of metabolic disease, has not been studied.

DETAILED DESCRIPTION:
This study was conducted in specific villages and hamlets that were randomly selected by multi-stage random cluster sampling in 2 provinces. The investigators randomly selected 36 villages (18 villages in each provinces) by using probability proportional to size cluster sampling to admit the total 360 women who met the criteria and consented. While Bifidobacterium, Advanced Glycation End Products (AGE) and lipid profile were examined in a subgroup of 120 participants from each province (n=240).

Field enumerators were trained to standardize 24 hours food recall, food frequency questionnaire for 1 month back, and for stool sampling technique procedure.

Anthropometric measurement was performed by performing weight and height measurement. Fasting blood sampling and fecal Bifidobacterium examination were done in collaboration with professional laboratories. Hemoglobin was assessed by using hemocue. Lipid profile was quantified using calorimetric method, fasting blood glucose (FBG) was quantified using enzymatic colorimetric method glucose oxidase - phenol aminophenazone, HbA1c was using high performance liquid chromatography (HPLC) hexokinase, malondialdehyde level was quantified using will's spectrophotometry, blood advance glycation end products was done by using enzyme linked immunosorbent assay (ELISA), carboxymethyl lysine plasma was done by ultra performance liquid chromatography-tandem mass spectometry (UPLC-MS/MS), and plasma tumor necrosis factor-alpha was done by ELISA. Fecal sample were collected in 2 pots, each contain 5-10 gram of stool, and store in cooler box (2-9 degree celcius) until sample was transported to laboratory as soon as possible to store in -80 degree celcius freezer.

ELIGIBILITY:
Inclusion Criteria:

* healthy reproductive women aged 19-50 years old
* having both parents from the same ethnicities (Minangkabau or Sundanese)
* willing to participate voluntarily signed a written informed-consent.

Exclusion Criteria:

* not being pregnant or lactating
* not having symptoms of gastrointestinal disturbance such as diarrhea, dysentery, constipation more than 3 days, and/or abdominal pain for the last 2 weeks
* not having nausea or vomiting or lost appetite for the last 2 days
* no history of malignancy
* not consuming antibiotics in the last 1 week before fecal collection
* not consuming alcohol more than 3 times a week

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Population represent mountainous and coastal areas (Tanah Datar and Padang Pariaman districts in West Sumatera for the Minangkabau ethnic group, and Tasikmalaya District in West Java for the Sundanese ethnic group), who are known to have differences in their traditional diets. These areas have agricultural fields, and the population of farmers and fishermen is above the regional average.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Dietary or nutritional intake | September - November 2016
  Usual dietary intake was done by using semi quantitative food frequency questionnaire for 1 month, and actual intake was done by nonconsecutive repeated 24-hour food recall (weekday and weekend). The investigators was analyse the dietary intake by Nutrisurvey 2007 software. Nutritional intake was reported as total daily intake (energy, macronutrients, and micronutrients). Energy intake is showed in kkal/day. Macronutrients include carbohydrate, protein, fat, and fiber intake are showed in gram/day. Micronutrients include vitamins and minerals are showed in gram/milligram/microgram per day. The value of nutrient intake are very diverse from 0 to high intake.

SECONDARY OUTCOMES:
Total fecal microbiota | September - December 2016
  Microbiota that examined in this study was total Bifidobacterium, quantified by real time-polymerase chain reaction, reported as log Bifidobacterium/gram feces. There is no official cut off for this measurement.
Weight | September - November 2016
  Body weight in kilograms
Height | September - November 2016
  Height in metres
Body mass index | September - November 2016
  Calculated from body weight divided by square of height, reported in kg/m2. Normal range 18.5-22.9 kg/m2.
Obesity | September - November 2016
  Classified using body mass index Asia Pacific standard. Score body mass index below 18.5 kg/m2 is underweight, 18.5-22.9 kg/m2 is normal range, 23-24.9 kg/m2 is overweight, 25-29.9 kg/m2 is obese 1, higher than 30 kg/m2 is obese 2
Waist circumference | September - November 2016
  Waist circumference in centimetres. Normal value is below 80 centimetres for women.
Hip circumference | September - November 2016
  Hip circumference in centimetres
Hemoglobin level | September - November 2016
  Blood hemoglobin was assessed by hemocue, reported in gram/decilitre. Normal value for blood hemoglobin is 12-15.5 gram/decilitre.
HbA1c | September - November 2016
  HbA1c was quantified using high performance liquid chromatography (HPLC) hexokinase, reported in %. Normal value is 4%-5.6%. Score 5.7%-6.4% means high risk of diabetes. Score 6.5% or higher for diagnose diabetes.
Lipid profile | September - November 2016
  Blood lipid profile was quantified using calorimetric method, reported as cholesterol total (normal value is less than 200 milligrams/decilitre)/ low density lipoprotein cholesterol (normal value is less than 100 milligrams/decilitre)/ high density lipoprotein cholesterol (normal value is higher than 40 milligrams/decilitre)/ triglyceride (normal value is less than 150 milligrams/decilitres).
Fasting blood glucose | September - November 2016
  Fasting blood glucose was quantified using enzymatic colorimetric method glucose oxidase - phenol aminophenazone. Normal value is less than 100 milligrams/decilitre.
Malondialdehyde (MDA) level | September - November 2016
  Blood MDA was quantified using spectrophotometry, reported in micromol/litre. There is no official cut off for this measurement.
Total advanced glycation end products (AGE) | September - December 2016
  Blood AGE was quantified by using enzyme linked immunosorbent assay (ELISA), reported in kilo unit/millilitre. There is no official cut off for this measurement.
Plasma carboxymethyl lysine (CML) | July - December 2017
  Plasma CML was quantified by ultra performance liquid chromatography-tandem mass spectometry (UPLC-MS/MS), reported in nanograms/millilitre. There is no official cut off for this measurement.
Tumor necrosis factor-alfa (TNF-alfa) | July - December 2017
  Plasma tumor necrosis factor-alpha was done by ELISA, reported in IU/millilitre. There is no official cut off for this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, Principal Investigator — Indonesia University

IPD SHARING:
Plan to Share IPD: No